CLINICAL TRIAL: NCT00513461
Title: A Phase II, Randomized, Controlled Trial of The Safety and Efficacy of S-Adenosyl-L-Methionine Disulphate P-Toluene-Sulfonate (SAMe) in Reducing Serum Alpha-Fetoprotein (AFP) in Patients With Hepatitis C and Moderately Elevated AFP
Brief Title: Liver Cancer Prevention Trial in Patients With Chronic Hep C Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chao Family Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Chao Family Comprehensive Cancer Center, Cancer Center, University of California, Irvine
Organization: University of California, Irvine (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UCI 06-07 / NCI-2009-00897; N01CN35160 (NIH); CDR0000558657 (Registry Identifier: PDQ (Physician Data Query)); UCI04-3-01 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Results first posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Adult Primary Liver Cancer; Hepatitis C Infection
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis C | interventions — Immunoenzyme Techniques; Chromatography, High Pressure Liquid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (SAMe) (Experimental): Patients receive SAMe PO QD for weeks 1-4, PO BID for weeks 5-8, and PO TID for weeks 9-24 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: S-adenosyl-L-methionine disulfate p-toluene-sulfonate; Other: laboratory biomarker analysis; Other: immunoenzyme technique; Other: high performance liquid chromatography
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO QD for weeks 1-4, PO BID for weeks 5-8, and PO TID for weeks 9-24 in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: placebo; Other: laboratory biomarker analysis; Other: immunoenzyme technique; Other: high performance liquid chromatography

INTERVENTIONS:
Drug: S-adenosyl-L-methionine disulfate p-toluene-sulfonate — Given PO
  Other Names: SAMe disulfate p-toluene-sulfonate
  Arms: Arm I (SAMe)
Other: placebo — Given PO
  Other Names: PLCB
  Arms: Arm II (placebo)
Other: laboratory biomarker analysis — Correlative studies
Other: immunoenzyme technique — Correlative studies
  Other Names: immunoenzyme techniques
Other: high performance liquid chromatography — Correlative studies
  Other Names: HPLC

SUMMARY:
This randomized phase II trial studies how well S-Adenosyl-L-Methionine Disulphate P-Toluene-Sulfonate (SAMe) works compared to a placebo in preventing liver cancer in patients with chronic hepatitis C infection. Chemoprevention is the use of certain drugs to keep cancer from forming. The use of SAMe may keep cancer from forming in patients with advanced liver disease

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether treatment with SAMe for 24 weeks reduces serum level of alpha-fetoprotein (AFP) in patients with advanced liver disease due to chronic hepatitis C.

SECONDARY OBJECTIVE:

I. To determine whether treatment with SAMe for 24 weeks reduces serum levels of des-gamma carboxyprothrombin (DCP) and alpha-fetoprotein-L3 (AFP-L3) in patients with advanced liver disease due to chronic hepatitis C (hepatocellular carcinoma tumor markers).

II. To determine whether treatment with SAMe for 24 weeks alters biochemical markers of liver disease (e.g., serum alanine aminotransferase [ALT], aspartate aminotransferase [AST], albumin, or bilirubin, etc.) and hepatitis C viral load in patients with advanced liver disease due to chronic hepatitis C (hepatitis C liver disease).

III. To determine whether treatment with SAMe for 24 weeks reduces serum levels of tumor necrosis factor-alpha (TNF-alpha), plasma levels of malondialdehyde (MDA), 4-hydroxynonenal (4-HNE) and urine levels of F2-isoprostane in patients with advanced liver disease due to chronic hepatitis C (oxidative stress).

IV. To determine whether treatment with SAMe for 24 weeks reduces plasma levels of methionine and homocysteine and increases plasma glutathione (GSH) and SAMe in patients with advanced liver disease due to chronic hepatitis C (SAMe metabolites).

V. To determine the safety, tolerability and quality of life of SAMe treatment (up to 2,400 mg/day) for 24 weeks in patients with advanced liver disease due to chronic hepatitis C.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive SAMe orally (PO) twice daily (BID) for 24 weeks in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive placebo PO once daily (QD) for weeks 1-4, PO BID for weeks 5-8, and PO three times daily (TID) for weeks 9-24 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C infection diagnosed by presence of hepatitis C ribonucleic acid (RNA) in serum by test of hepatitis C virus (HCV) RNA
* No significant alcohol use (7 or fewer drinks per week) for the past 12 months
* Serum AFP (at screening) between 15 and 100 ng/mL (15 ng/mL =< AFP =< 100 ng/mL) as measured by the Bayer Advai Centaur chemiluminescence system OR Serum AFP between 10 and 100 ng/mL (10 ng/mL =< AFP =<100 ng/mL) as measured by Diagnostic Products Corporation Immulite assay system OR AFP between 12 and 100 ng/mL (12 ng/mL =< AFP =< 100 ng/mL) as measured by Ortho ECiQ assay system
* Evidence of advanced liver disease based on one or more of the following:
* Platelet count less than 150,000/mm^3
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ratio > 0.75
* Liver biopsy demonstrating bridging fibrosis or cirrhosis
* No treatment with interferon (recombinant interferon alfa), peginterferon (PEG-interferon alfa-2b), or ribavirin for at least 4 months, and not anticipated to start specific treatment for hepatitis C during the study (30 weeks)
* Ultrasound (or adequate computed tomography [CT] or magnetic resonance imaging [MRI]) examination of the liver within 6 months prior to randomization revealing no masses in the liver suggestive of hepatocellular carcinoma
* Willing to refrain from consuming over-the-counter SAMe and vitamin pills containing B-vitamins while participating in this study (30 weeks)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Leukocytes > 1,000/ mm^3
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Liver disease other than from hepatitis C (e.g., hepatitis B, hemochromatosis, fat in more than 33% of hepatocytes, if liver biopsy has been performed., etc.); subjects with a past history of alcohol use can be enrolled into the study provided they have consumed less than 7 drinks/week for the past 12 months
* Evidence of mass in liver by radiologic examination that is suggestive of hepatocellular carcinoma within 6 months prior to randomization
* Model for End-Stage Liver Disease (MELD) score greater than 15 within 60 days prior to enrollment
* Ascites which is clinically detectable
* Use of SAMe during 4 months prior to randomization
* Hospitalization within the past 5 years for mania or for bipolar disease
* Concurrent use of monoamine oxidase inhibitors (MAO) or other drugs that increase the concentration of serotonin
* Participants may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to SAMe
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Children are excluded from this study but will be eligible for future pediatric trials, if applicable
* Pregnant women are excluded from this study; serum pregnancy must be performed and be negative in all women of child bearing potential within 2 weeks prior to enrollment; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with SAMe, breastfeeding should be discontinued if the mother is treated with SAMe
* Subjects with any medical psychosocial condition that, in the opinion of the investigator, could jeopardize the subject's participation in and compliance with the study criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2007-10; Primary Completion 2012-08 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Hoefs, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (5):
- United States (5):
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - Veterans Administration Long Beach Medical Center, Long Beach, California
  - Veterans Administration Los Angeles Healthcare System, Los Angeles, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California At San Diego, San Diego, California

REFERENCES:
- [Result] Morgan TR, Osann K, Bottiglieri T, Pimstone N, Hoefs JC, Hu KQ, Hassanein T, Boyer TD, Kong L, Chen WP, Richmond E, Gonzalez R, Rodriguez LM, Meyskens FL. A Phase II Randomized, Controlled Trial of S-Adenosylmethionine in Reducing Serum alpha-Fetoprotein in Patients with Hepatitis C Cirrhosis and Elevated AFP. Cancer Prev Res (Phila). 2015 Sep;8(9):864-72. doi: 10.1158/1940-6207.CAPR-15-0029. Epub 2015 Jun 30. PMID 26130251

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (SAMe) | Arm II (Placebo)
Started | 57 | 53
Completed | 44 | 43
Not Completed | 13 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (SAMe) | Arm II (Placebo) | Total
Number analyzed (Participants) | 57 | 53 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (4.9) | 57.2 (5.8) | 57.88 (5.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 48 | 47 | 95

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum AFP Levels
Description: Measured using an Food and Drug Administration (FDA)-approved assay. Mean change over time for the SAMe and placebo groups will be estimated. Differences in the change over time between the treated and control groups will be tested using a two-group repeated measures analysis of variance model.
Time Frame: Baseline to week 24
Population: All subjects who completed the week 24 visit as planned were included in the data anlysis. The number of subjects in each analysis differed slightly because the number of subjects with data at both time points (i.e., week 0 and week 24) varied depending on the outcome measured.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm I (SAMe) | Arm II (Placebo)
Number analyzed (Participants) | 43 | 40
ng/mL | -1.928 (20.304) | 5.855 (29.207)
Statistical Analysis 1: Comparison: Arm I (SAMe) vs Arm II (Placebo); Test type: Superiority; p = 0.160, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 7.78

2. Secondary Outcome: Treatment-related Changes in Serum DCP for Hepatocellular Carcinoma
Description: To determine whether treatment with SAMe for 24 weeks reduces serum levels of des-gamma carboxyprothrombin (DCP) in patients with advanced liver disease due to chronic hepatitis C (hepatocellular carcinoma tumor markers).
Time Frame: Baseline to week 24
Population: All subjects who completed the week 24 visit as planned were included in the data analysis. The number of subjects in each analysis differed slightly because the number of subjects with data at both time points (i.e., week 0 and week 24) varied depending on the outcome measured.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm I (SAMe) | Arm II (Placebo)
Number analyzed (Participants) | 27 | 26
ng/mL | 0.259 (0.976) | 0.647 (1.491)

3. Secondary Outcome: Treatment-related Changes in Serum AFP-L3 (Expressed as the Percentage of Total AFTP) for Hepatocellular Carcinoma
Description: AFP-L3 assay will be performed by Wako Laboratories using their LiBASys platform.
Time Frame: Baseline to week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of AFP-L3/AFP
Arm/Group | Arm I (SAMe) | Arm II (Placebo)
Number analyzed (Participants) | 27 | 26
percentage of AFP-L3/AFP | 0.144 (1.146) | 0.335 (3.486)

4. Secondary Outcome: SAMe
Description: Change in SAMe levels
Time Frame: Baseline to week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Arm I (SAMe) | Arm II (Placebo)
Number analyzed (Participants) | 43 | 41
nmol/L | 414.242 (744.373) | -9.085 (54.621)

5. Secondary Outcome: Change in SAMe Metabolites - S-adenosylhomocysteine (SAH)
Description: S-adenosylhomocysteine (SAH)
Time Frame: Baseline to week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Arm I (SAMe) | Arm II (Placebo)
Number analyzed (Participants) | 43 | 41
nmol/L | 16.326 (28.212) | -3.456 (13.104)

6. Secondary Outcome: Change in SAMe Metabolites - Methionine
Description: Methionine will be measured using HPLC with fluorescence detection.
Time Frame: Baseline to week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Arm I (SAMe) | Arm II (Placebo)
Number analyzed (Participants) | 43 | 41
µmol/L | 0.421 (18.794) | -2.894 (23.669)

7. Secondary Outcome: Change in SAMe Metabolites - Total Homocysteine (tHcy)
Description: Total homocysteine (tHcy)
Time Frame: Baseline to week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Arm I (SAMe) | Arm II (Placebo)
Number analyzed (Participants) | 43 | 41
µmol/L | 0.266 (2.394) | -0.677 (2.478)

8. Secondary Outcome: Change in SAMe Metabolites - Plasma GSH
Description: Plasma GSH will be measured using HPLC with fluorescence detection.
Time Frame: Baseline to week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Arm I (SAMe) | Arm II (Placebo)
Number analyzed (Participants) | 43 | 41
µmol/L | 0.455 (1.425) | 0.285 (1.23)

9. Secondary Outcome: Change in SAMe Metabolites - Malondialdehyde (MDA)
Description: malondialdehyde
Time Frame: Baseline to week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Arm I (SAMe) | Arm II (Placebo)
Number analyzed (Participants) | 43 | 41
µmol/L | -0.007 (0.848) | -0.002 (1.162)

10. Secondary Outcome: Change in SAMe Metabolites - 4-hydroxynonenal (4-HNE)
Description: Serum marker of oxidative stress. One mechanism by which SAMe is hypothesized to be beneficial is by reducing oxidative stress.
Time Frame: Baseline to week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Arm I (SAMe) | Arm II (Placebo)
Number analyzed (Participants) | 43 | 41
µg/mL | -0.185 (0.716) | -0.032 (0.448)

11. Secondary Outcome: Change in Markers of Liver Disease - AST
Description: AST measurements will be performed in a College of American Pathologists (CAP)-certified lab using FDA-approved assays.
Time Frame: Baseline to week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Arm I (SAMe) | Arm II (Placebo)
Number analyzed (Participants) | 44 | 43
IU/L | -0.755 (37.531) | 1.723 (40.709)

12. Secondary Outcome: Change in Markers of Liver Disease - ALT
Description: ALT measurements will be performed in a College of American Pathologists (CAP)-certified lab using FDA-approved assays.
Time Frame: Baseline to week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Arm I (SAMe) | Arm II (Placebo)
Number analyzed (Participants) | 44 | 43
IU/L | -9.548 (34.786) | 0.019 (41.165)

13. Secondary Outcome: HCV RNA
Description: Change in HCV RNA levels. Serum level of HVC RNA was measured using COBAS TaqMan HCV test (Roche Molecular Systems).
Time Frame: Baseline to week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Arm I (SAMe) | Arm II (Placebo)
Number analyzed (Participants) | 36 | 35
IU/mL | -259327.69 (3084015.42) | -19968.89 (2425010.48)

14. Secondary Outcome: Changes in Quality of Life - Physical Score
Description: Change from Baseline to Week 24 in Quality of life as as assessed with Short Form (SF)-36 Physical Component Scores. Measured quality of life using the SF-36, a widely used and general questionnaire of quality of life. Possible scores range from 0 and 100. High scores reflect good QOL and low scores reflect bad QOL. Change in QOL = (Week 24 score - Baseline score).
Time Frame: Baseline to week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (SAMe) | Arm II (Placebo)
Number analyzed (Participants) | 43 | 43
units on a scale | -0.4 (11.73) | 0.03 (13.6)
Statistical Analysis 1: Comparison: Arm I (SAMe) vs Arm II (Placebo); Test type: Superiority; p = 0.878, Two-Group t-test; Mean Difference (Net) = 0.43

15. Secondary Outcome: Changes in Quality of Life - Mental Score
Description: Change from Baseline to Week 24 in Quality of life as as assessed with Short Form (SF)-36 Mental Component Scores. Measured quality of life using the SF-36, a widely used and general questionnaire of quality of life. Possible scores range from 0 and 100. High scores reflect good QOL and low scores reflect bad QOL. Change = (Week 24 score - Baseline score).
Time Frame: Baseline to week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Arm I (SAMe) | Arm II (Placebo)
Number analyzed (Participants) | 43 | 43
scores on a scale | 0.83 (15.06) | -2.83 (11.76)
Statistical Analysis 1: Comparison: Arm I (SAMe) vs Arm II (Placebo); Test type: Superiority; p = 0.212, Two-Group t-test; Mean Difference (Net) = -3.66

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 30 weeks.
Arm/Group | Arm I (SAMe) | Arm II (Placebo)
Serious Adverse Events (participants affected / at risk) | 5/57 | 3/53
Other Adverse Events (participants affected / at risk) | 51/57 | 46/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (SAMe) (N=57) | Arm II (Placebo) (N=53)
ABDOMINAL CELLULITIS (Infections and infestations) | 0 (0) | 1 (1)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN.STATUS POST SPLENIC ARTERY EMBOLIZATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
ANGIOPLASTY OF LEFT HYPOGASTRIC ARTERY, EXTERNAL ILIAC STENT PLACEMENT FOR LEFT LEG (Vascular disorders) | 0 (0) | 1 (1)
HEPATOCELLULAR CARCINOMA (Hepatobiliary disorders) | 0 (0) | 1 (1)
LEFT THIGH ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
NEPHROTIC SYNDROME (Renal and urinary disorders) | 1 (1) | 0 (0)
NON-ST ELEVATION MIOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
SMALL BOWEL INFLAMATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
SPLENOMEGALY SECONDARY TO PORTAL HYPERTENSION (Hepatobiliary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (SAMe) (N=57) | Arm II (Placebo) (N=53)
ABDOMINAL CRAMPS (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 (1) | 0 (0)
ALLERGIC RHINITIS (Immune system disorders) | 0 (0) | 1 (1)
ANAL IRRITATION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 3 (3) | 0 (0)
ARTHRITIS PAIN, KNEES (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ARTHRITIS PAIN, LOWER BACK (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ASCITES (Gastrointestinal disorders) | 1 (1) | 2 (2)
BAD GAS (Gastrointestinal disorders) | 1 (1) | 1 (1)
BLACK OUT (Nervous system disorders) | 0 (0) | 1 (1)
BLEEDING ESPHAGEAL VARICES (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
BLOOD IN STOOLS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
BLURRED VISION (Eye disorders) | 0 (0) | 1 (1)
BORDERLINE DIABETES (Endocrine disorders) | 1 (1) | 0 (0)
BREAST TENDERNESS (Reproductive system and breast disorders) | 1 (1) | 0 (0)
BROKEN TOOTH-UNCOMPLICATED (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
BRUISING R LEG (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
CELLULITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
CHEST CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
CHILLS (General disorders) | 1 (1) | 0 (0)
CHRONIC ASCITES (Gastrointestinal disorders) | 0 (0) | 1 (1)
CHRONIC GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
CLICKING SOUND IN THE HEAD (Ear and labyrinth disorders) | 1 (1) | 0 (0)
COLD (General disorders) | 4 (5) | 2 (2)
COMMON COLD (General disorders) | 1 (1) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 12 (17) | 5 (6)
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
CYST ON PATELLA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DARK COLORED URINE (Renal and urinary disorders) | 0 (0) | 1 (1)
DECREASED INSOMNIA (Psychiatric disorders) | 1 (1) | 0 (0)
DENTAL IMPLANT SURGERY (Gastrointestinal disorders) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 1 (1)
DIABETES MELLITUS (Endocrine disorders) | 0 (0) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 20 (31) | 13 (17)
DIARRHEA 4-6 STOOLS/DAY (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIFFUSE ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
DISLOCATION OF LEFT SHOULDER (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 5 (6) | 4 (6)
DRY MOUTH (Gastrointestinal disorders) | 10 (10) | 12 (13)
DRY MOUTH/SALIVARY GLAND (Gastrointestinal disorders) | 1 (1) | 0 (0)
DRYNESS OF MOUTH (Gastrointestinal disorders) | 1 (1) | 0 (0)
EAR PAIN (Ear and labyrinth disorders) | 0 (0) | 1 (1)
EARS RINGING (Ear and labyrinth disorders) | 0 (0) | 1 (1)
ELEVATED AFP (Renal and urinary disorders) | 0 (0) | 1 (1)
ELEVATED CREATININE (Investigations) | 1 (1) | 0 (0)
ELEVATED INR (Investigations) | 1 (1) | 0 (0)
EXTRA GAS FLATULENCE (Gastrointestinal disorders) | 0 (0) | 1 (1)
EYE PAIN (Eye disorders) | 0 (0) | 1 (1)
EYES HURT (Eye disorders) | 1 (1) | 0 (0)
FACIAL SWELLING OF ALLERGIC ORIGIN (Immune system disorders) | 1 (1) | 0 (0)
FALL, HIP AND BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 15 (19) | 9 (11)
FEET AND LEGS CRAMPS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
FEVER (General disorders) | 1 (1) | 1 (1)
FLATULENCE (Gastrointestinal disorders) | 19 (22) | 22 (25)
FLU (General disorders) | 1 (1) | 0 (0)
FLU-LIKE SYMPTOMS (General disorders) | 0 (0) | 4 (4)
FOOD POISONING (Gastrointestinal disorders) | 2 (2) | 0 (0)
FORGETFULNESS (Nervous system disorders) | 0 (0) | 1 (1)
FRACTURE 5TH R METACARPAL (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
GAS-FLATULENCE (Gastrointestinal disorders) | 1 (1) | 1 (1)
GI CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
GUM BLEEDING (Gastrointestinal disorders) | 0 (0) | 1 (1)
HAIR LOSS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
HAPPIER (Psychiatric disorders) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 13 (16) | 11 (13)
HEADACHE-SINUS (Nervous system disorders) | 0 (0) | 1 (1)
HEARTBURN (Gastrointestinal disorders) | 7 (9) | 4 (4)
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 1 (1)
HOT FLUSHES (Endocrine disorders) | 1 (1) | 0 (0)
HUNGRIER (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
HYPERSOMNIA (Psychiatric disorders) | 2 (2) | 0 (0)
HYPOKALEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
INCREASE IN FLATULENCE (Gastrointestinal disorders) | 1 (1) | 0 (0)
INCREASE NUMBER OF STOOLS (Gastrointestinal disorders) | 1 (1) | 0 (0)
INCREASE PEE (Renal and urinary disorders) | 0 (0) | 1 (1)
INCREASED DIARRHEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
INCREASED FLATULENCE (Gastrointestinal disorders) | 0 (0) | 1 (1)
INCREASED STOMACH PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
INCREASED SWEATING (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
INCREASED URINATION (Renal and urinary disorders) | 12 (13) | 9 (10)
INFECTED SEBACEOUS CYST R. AXILA (Infections and infestations) | 1 (1) | 0 (0)
INSOMNIA (Psychiatric disorders) | 9 (11) | 8 (9)
INTERMITTENT HEADACHE (Nervous system disorders) | 1 (1) | 1 (1)
INTESTINAL FLU (Gastrointestinal disorders) | 1 (1) | 0 (0)
INVOLUNTARY MOVEMENT (Nervous system disorders) | 1 (1) | 1 (1)
IRRITABILITY (Psychiatric disorders) | 0 (0) | 1 (1)
ITCHINESS ALL OVER THE BODY (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
ITCHING (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
JOINT PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
KNEE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
LEFT LEG VASCULAR CLAUDICATION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
LEFT SIDE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
LEG CRAMPS (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
LOWER BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
LOWER BACK SURGERY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
LOWER BACKACHE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
LOWER EXTREMITY EDEMA (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
MACULOPAPULAR RASH ON TORSO (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
MANIA (Psychiatric disorders) | 1 (1) | 2 (5)
MEMORY LOSS (Nervous system disorders) | 0 (0) | 1 (1)
MILD RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
MOOD ALTERATION (Psychiatric disorders) | 2 (7) | 2 (2)
MOOD ALTERATION DEPRESSION (Psychiatric disorders) | 1 (2) | 0 (0)
MOOD ALTERATION-ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0)
MOOD ALTERATION-HAPPY (Psychiatric disorders) | 1 (1) | 0 (0)
MOOD ALTERATION:ANXIETY (Psychiatric disorders) | 0 (0) | 1 (1)
MUSCLE CRAMPS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
MUSCLE CRAMPS OF BOTH LEGS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCLE MOVEMENT (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL PAIN (NECK) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 18 (20) | 7 (8)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
NOSE BLEEDING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OLECRANON BURSITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN IN BOTH HANDS AND FEET (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN IN KNEE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN LEFT SIDE OF CHEST (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN ON ANKLE JOINTS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN ON HIP (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN ON KNEE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PINCHED NERVE (Nervous system disorders) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
QUEASINESS (Gastrointestinal disorders) | 0 (0) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
RASH ON BOTH ARMS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RASH ON EXTREMETIES (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RESPIRATORY TRACT INFECTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESTLESSNESS (Psychiatric disorders) | 0 (0) | 1 (1)
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
SINUS PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SINUSITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
SKIN RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
SPRAINED ANKLE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
STIFF NECK (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
STIFFNESS OF JOINTS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
STOMACH ACHE (Gastrointestinal disorders) | 1 (1) | 0 (0)
STOMACH CRAMPS (Gastrointestinal disorders) | 1 (3) | 0 (0)
STOMACH FLU (Gastrointestinal disorders) | 0 (0) | 1 (1)
STOMACH PAIN (Gastrointestinal disorders) | 21 (28) | 9 (10)
SWEATING (Skin and subcutaneous tissue disorders) | 5 (5) | 6 (9)
SWEATING "NIGHT" (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SWELLING OF ANKLES (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
TICS (Nervous system disorders) | 0 (0) | 1 (1)
TINNITUS (Ear and labyrinth disorders) | 0 (0) | 1 (1)
TIREDNESS FATIGUE (General disorders) | 0 (0) | 1 (1)
TOOTH EXTRACTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 1 (1) | 0 (0)
ULCERATION OF THE LIP (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
UPSET STOMACH (Gastrointestinal disorders) | 0 (0) | 1 (1)
URINE ODOR (Renal and urinary disorders) | 0 (0) | 1 (1)
VAGINAL IRRITATION (Reproductive system and breast disorders) | 1 (1) | 0 (0)
VAGINAL YEAST INFECTION (Infections and infestations) | 0 (0) | 1 (1)
VIRAL INFECTION INCLUDING COUGHING (Infections and infestations) | 1 (1) | 0 (0)
VITAMIN D DEFICIENCY (Investigations) | 0 (0) | 1 (1)
VIVID DREAMS (Psychiatric disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 5 (6) | 4 (4)
WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
WEIGHT GAIN (Investigations) | 1 (1) | 0 (0)
WORSENING OF ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0)
WORSENING OF BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
WORSENING OF BASELINE DIABETES MELLITUS (Endocrine disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less